CLINICAL TRIAL: NCT00894140
Title: A Non-comparative, Two Centre, EN540, RSA, Pilot Study to Evaluate the Stability, Efficacy and Safety of the Silent Hip Prosthesis in Primary Total Hip Replacement
Brief Title: Study to Assess the Stability, Efficacy and Safety of the Silent™ Hip Prosthesis in Primary Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy International (Industry)
Collaborators: Johnson and Johnson Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT01/27
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis
Keywords: Hip; Cementless; Conservative
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy Silent™ Hip femoral prosthesis (Other): A short cementless, femoral component for use in total hip arthroplasty
  Interventions: Device: DePuy Silent™ Hip femoral prosthesis

INTERVENTIONS:
Device: DePuy Silent™ Hip femoral prosthesis — A short cementless, femoral component for use in total hip arthroplasty

SUMMARY:
The purpose of this study is to determine if the Silent™ hip, when used as part of an artificial hip joint, is stable and effective in treatment of patients with joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical, standard and special x-rays (RSA) to allow the position of the Silent Hip within the bone to be accurately monitored.

DETAILED DESCRIPTION:
The Primary Objective of this study was to evaluate the short-term stability of the Silent Hip, implanted using a manual or navigated technique, using radiostereometric analysis (RSA). The study was also intended to provide the clinical data necessary to demonstrate conformance with the essential requirements of the Medical Device Directive. Secondary objectives were to determine the efficacy of the Silent™ Hip femoral prosthesis from a clinical and radiological prospective, to assess the safety of the device and to evaluate the impact of the procedure on the Subjects' Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged between 25 and 65 years inclusive.
2. Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
3. Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
4. Subjects with non-inflammatory osteoarthritis of the hip who require a primary total hip replacement.

Exclusion Criteria:

1. Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
2. Women who are pregnant.
3. Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
4. Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).
5. Subjects who are currently involved in any injury litigation claims.
6. Subjects who have osteonecrosis of the femoral neck
7. Subjects who have an existing contralateral hip, ankle or knee replacement or an ipsilateral knee or ankle replacement or any metal implant in the lower lumber spine (navigated cases only).
8. Subjects who are greater than 90kg in weight.
9. Subject who have a CCD angle of the anatomical femur less than 125˚
10. Subjects with significant bone loss or gross deformity in the region of the neck of the femur as identified on the pre-operative radiographs, where in the Investigator's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the prosthesis.
11. Subjects with a Charnley C classification.
12. Subjects with an active local or systemic infection.
13. Subjects with loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the arthroplasty procedure unjustified.
14. Subjects with Paget's disease
15. Subjects who still plan in the future to have children.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-01; Primary Completion 2004-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The translational and rotational movements of the Silent™ hip in the 3 dimensions from the baseline position (determined from the 7 day post-operative RSA x-rays) to the 1 year follow-up visit. | 1year post-surgery

SECONDARY OUTCOMES:
Kaplan Meier survivorship of the Silent Hip prosthesis in terms of revision and radiological aseptic loosening | 1 year
Difference demonstrated between pre-op and 5 year Harris Hip Score | 5 years post surgery
Difference demonstrated between pre-op and 5 year Oxford Hip Score | 5years post surgery
Incidence of radiological signs on the post-operative x-rays | 3 months post surgery
Difference demonstrated between pre-op and 10 year Harris Hip Score | 10 years post surgery
Difference demonstrated between pre-op and 10 year Oxford Hip Score | 10 years post surgery
Incidence of radiological signs on the post-operative x-rays | 6 months post surgery
Incidence of radiological signs on the post-operative x-rays | 1 year post surgery
Incidence of radiological signs on the post-operative x-rays | 18 months post surgery
Incidence of radiological signs on the post-operative x-rays | 2 years post surgery
Incidence of radiological signs on the post-operative x-rays | 5 years post surgery
Incidence of radiological signs on the post-operative x-rays | 10 years post surgery
Kaplan Meier survivorship of the Silent Hip prosthesis in terms of revision and radiological aseptic loosening | 2 years
Kaplan Meier survivorship of the Silent Hip prosthesis in terms of revision and radiological aseptic loosening | 5 years
Kaplan Meier survivorship of the Silent Hip prosthesis in terms of revision and radiological aseptic loosening | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammy ODell, BS, Study Chair — DePuy International
Locations (2):
- Sydney Adventist Hospital, Sydney, Australia
- General Hospital Eilbek, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No